CLINICAL TRIAL: NCT01534858
Title: A Prospective, Descriptive Cohort Study With Prontosan® Wound Gel X in Partial and Full Thickness Burns Requiring Split Thickness Skin Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Ltd. Centre of Excellence Infection Control (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OPM-O-H-1102
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2015-09

CONDITIONS: Burns
Keywords: polyhexanide, polihexanide, PHMB, Prontosan, burns, wounds
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Partial and full thickness burns with split thickness grafts (Experimental)
  Interventions: Device: Prontosan Wound Gel X

INTERVENTIONS:
Device: Prontosan Wound Gel X — Prontasan Wound Gel X will be applied topically as a thin layer to the entire grafted area immediately after transplant and with each dressing change.
  Other Names: polihexanide and betaine containing hydrogel

SUMMARY:
The purpose of this study is to evaluate the healing of split thickness skin grafts when treated with Prontosan® Wound Gel X in patients with partial and full thickness skin burns.

ELIGIBILITY:
Inclusion Criteria:

* Partial of full thickness burns requiring split thickness grafts
* Target burn wound size 10cm2-1000cm2
* Age ≥ 18 years
* Ability to read, write and speak German.
* Provision of voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent approved by the Institutional Ethics Committee (IEC) prior to all evaluations. Informed consent will be obtained from the patient or by a legal representative if the patient is not able/competent to consent. In this case, informed consent will be also obtained by the patient when he/she regains competence.
* Women of child bearing potential must test negative on standard urine pregnancy test and must agree to practice appropriate contraceptive methods for the duration of the study (e. g. oral contraceptive, IUD, intra-muscular contraceptive, abstinence).

Exclusion Criteria:

* Target wound has exposed hyaline cartilage
* Connective tissue disorder
* Previous skin graft failure at target wound site
* Total burn surface area ≥ 70%
* Infected target wound
* Immunosuppression therapy
* Chronic hemodialysis
* Steroid use
* Diabetes (Type I)
* Allergy or sensitivity to any of the ingredients in Prontosan® Wound Gel X
* Allergy or sensitivity to chlorhexidine
* Pregnancy
* Simultaneous participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Graft neo-epithelisation | 29 days
Time to complete epithelization | 29 days
Wound infection | 29 days
Need for re-operation of target wound site | 29 days

SECONDARY OUTCOMES:
Pain | 29 days
Pruritis | 29 days
Erythema | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Daigeler, Prof., Principal Investigator — Berufsgenossenschaftliches Unfallklinikum Bergmannsheil Bochum; Jurij Kiefer, Dr., Principal Investigator — Berufsgenossenschaftliche Unfallklinik Ludwigshafen; Adrian Dragu, PD Dr. med., Principal Investigator — Klinikum St. Georg Leipzig
Locations (3):
- Germany (3):
  - Berufsgenossenschaftliche Unfallklinik Ludwigshafen, Ludwigshafen, Baden-Wurttemberg
  - Berufsgenossenschaftliches Unfallklinikum Bergmannsheil, Bochum
  - Klinikum St. Georg, Leipzig

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/29668985